CLINICAL TRIAL: NCT00937404
Title: An Open-label Primary Vaccination Study to Assess the Safety and Reactogenicity of GlaxoSmithKline Biologicals' Inactivated Poliomyelitis Vaccine Poliorix Administered as a Three-dose Primary Vaccination Course at 2, 3 and 4 Months of Age in Healthy Infants in China.
Brief Title: Safety and Reactogenicity of GSK Biologicals' Inactivated Poliomyelitis Vaccine (IPV) (Poliorix) in Infants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 112581
Record Dates: First submitted 2009-07-09; First posted 2009-07-13 (Estimated); Results first posted 2018-12-17 (Actual); Last update posted 2018-12-17 (Actual); Status verified 2018-05

CONDITIONS: Poliomyelitis
Keywords: IPV
MeSH Terms: conditions — Poliomyelitis

ARMS (1):
- IPV Group (Experimental): Healthy male or female subjects between, and including, 60 and 90 days of age at the time of the first vaccination, receive 3 doses of Poliorix at 2 (Study Day 0, Visit 1), 3 (Study Month 1, Visit 2) and 4 (Study Month 2, Visit 3) months of age, administered intramuscularly into the upper right side of the thigh.
  Interventions: Biological: Poliorix

INTERVENTIONS:
Biological: Poliorix — All subjects receive three doses of Poliorix vaccine, administered intramuscularly into the upper right side of the thigh.

SUMMARY:
The study will evaluate the safety and reactogenicity of Poliorix given as primary vaccination course to Chinese children at 2, 3 and 4 months of age.

ELIGIBILITY:
Inclusion Criteria:

* A male or female infant between, and including, 60 and 90 days of age at the time of the first vaccination.
* Born after a gestation period of 36 to 42 weeks inclusive.
* Subjects who the investigator believes that their parents/ guardians can and will comply with the requirements of the protocol should be enrolled in the study.
* Written informed consent obtained from the parent or guardian of the subject.
* Healthy subjects as established by medical history and clinical examination before entering into the study.

Exclusion Criteria:

* Use of any investigational or non-registered product other than the study vaccine(s) within 30 days preceding the first dose of study vaccine, or planned use during the study period.
* Chronic administration of immunosuppressants or other immune-modifying drugs since birth.
* Administration of immunoglobulins and/or any blood products since birth or planned administration during the study period.
* Administration of a vaccine not foreseen by the study protocol within 30 days prior to vaccination, or planned administration during the study period, with exception of DTP, Hib and/or hepatitis B vaccine(s).
* Concurrently participating in another clinical study, at any time during the study period, in which the subject has been or will be exposed to an investigational or a non-investigational product.
* Evidence of previous or intercurrent poliomyelitis disease or vaccination.
* History of seizures or progressive neurological disease.
* Any confirmed or suspected immunosuppressive or immunodeficient condition, based on medical history and physical examination.
* History of allergic disease or reactions likely to be exacerbated by any component of the vaccine(s).
* Major congenital defects or serious chronic illness. The following condition is temporary or self-limiting and a subject may be vaccinated once the condition has resolved and no other exclusion criteria are met:
* Current febrile illness or axillary temperature > 37.0 ºC or other moderate to severe illness within 24 hours of study vaccine administration.

Ages: 60 Days to 90 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 25 (Actual)
Dates: Start 2009-08-04 (Actual); Primary Completion 2009-11-13 (Actual); Study Completion 2009-11-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Wuzhou, Guangxi, China

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Derived] Li R, Li CG, Li Y, Liu Y, Zhao H, Chen X, Kuriyakose S, Van Der Meeren O, Hardt K, Hezareh M, Roy-Ghanta S. Primary and booster vaccination with an inactivated poliovirus vaccine (IPV) is immunogenic and well-tolerated in infants and toddlers in China. Vaccine. 2016 Mar 14;34(12):1436-43. doi: 10.1016/j.vaccine.2016.02.010. Epub 2016 Feb 9. PMID 26873055
- See also: Results for study 112581 can be found on the GSK Clinical Study Register — https://www.gsk-clinicalstudyregister.com/study/112581?search=study&b%22b''%22#rs
- Available data/document: Study Protocol: 112581 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 112581 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 112581 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 112581 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 112581 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 112581 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register

RESULTS

PARTICIPANT FLOW:
Groups:
- IPV Group: Healthy male or female subjects between, and including, 60 and 90 days of age at the time of the first vaccination, received 3 doses of Poliorix at 2 (Study Day 0, Visit 1), 3 (Study Month 1, Visit 2) and 4 (Study Month 2, Visit 3) months of age, administered intramuscularly into the upper right side of the thigh.
Period: Overall Study
Arm/Group | IPV Group
Started | 25
Completed | 23
Not Completed | 2
Not completed — Protocol Violation | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Arm/Group | IPV Group
Number analyzed (Participants) | 25
Age, Continuous [Mean (Standard Deviation); unit: Weeks] | 9.6 (1.38)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15
  Male | 10
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian-Chinese Heritage | 25

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects Reporting Solicited Local Symptoms
Description: Solicited local symptoms assessed were pain, redness and swelling. Any = occurrence of the symptom irrespective of intensity grade. Grade 3 pain = cried when limb was moved/spontaneously painful. Grade 3 redness/swelling = redness/swelling spreading beyond 30 millimetres (mm) of injection site.
Time Frame: During the 4-day follow-up period after each dose of study vaccine.
Population: Analysis was performed on the Total Vaccinated Cohort, which included all subjects with documented administration of at least one dose of the study vaccine.
Measure: Count of Participants; unit: Participants
Arm/Group | IPV Group
Number analyzed (Participants) | 25
Participants
  Any Pain, Dose 1 | 1
  Grade 3 Pain, Dose 1 | 0
  Any Redness, Dose 1 | 2
  Grade 3 Redness, Dose 1 | 0
  Any Swelling, Dose 1 | 1
  Grade 3 Swelling, Dose 1 | 0
  Any Pain, Dose 2: number analyzed (Participants) | 23
  Any Pain, Dose 2 | 2
  Grade 3 Pain, Dose 2: number analyzed (Participants) | 23
  Grade 3 Pain, Dose 2 | 0
  Any Redness, Dose 2: number analyzed (Participants) | 23
  Any Redness, Dose 2 | 1
  Grade 3 Redness, Dose 2: number analyzed (Participants) | 23
  Grade 3 Redness, Dose 2 | 0
  Any Swelling, Dose 2: number analyzed (Participants) | 23
  Any Swelling, Dose 2 | 1
  Grade 3 Swelling, Dose 2: number analyzed (Participants) | 23
  Grade 3 Swelling, Dose 2 | 0
  Any Pain, Dose 3: number analyzed (Participants) | 23
  Any Pain, Dose 3 | 1
  Grade 3 Pain, Dose 3: number analyzed (Participants) | 23
  Grade 3 Pain, Dose 3 | 0
  Any Redness, Dose 3: number analyzed (Participants) | 23
  Any Redness, Dose 3 | 0
  Grade 3 Redness, Dose 3: number analyzed (Participants) | 23
  Grade 3 Redness, Dose 3 | 0
  Any Swelling, Dose 3: number analyzed (Participants) | 23
  Any Swelling, Dose 3 | 0
  Grade 3 Swelling, Dose 3: number analyzed (Participants) | 23
  Grade 3 Swelling, Dose 3 | 0
  Any Pain, Across doses | 3
  Grade 3 Pain, Across doses | 0
  Any Redness, Across doses | 2
  Grade 3 Redness, Across doses | 0
  Any Swelling, Across doses | 2
  Grade 3 Swelling, Across doses | 0

2. Primary Outcome: Number of Subjects Reporting Solicited General Symptoms
Description: Assessed solicited general symptoms were drowsiness, irritability, loss of appetite and fever [defined as axillary temperature equal to or above (≥) 37.1 degrees Celsius (°C)]. Any = occurrence of symptom regardless of intensity grade of relationship to vaccination. Grade 3 drowsiness = drowsiness that prevented normal activity. Grade 3 irritability = crying that could not be comforted/prevented normal activity. Grade 3 loss of appetite = subject did not eat at all. Grade 3 fever = fever above (>) 39.0°C. Related = symptom assessed by the investigator as related to vaccination.
Time Frame: During the 4-day follow-up period after each dose of study vaccine.
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | IPV Group
Number analyzed (Participants) | 25
Participants
  Any Drowsiness, Dose 1 | 7
  Grade 3 Drowsiness, Dose 1 | 0
  Related Drowsiness, Dose 1 | 7
  Any Irritability, Dose 1 | 10
  Grade 3 Irritability, Dose 1 | 0
  Related Irritability, Dose 1 | 10
  Any Loss of appetite, Dose 1 | 7
  Grade 3 Loss of appetite, Dose 1 | 0
  Related Loss of appetite, Dose 1 | 7
  Any Fever, Dose 1 | 8
  Grade 3 Fever, Dose 1 | 0
  Related Fever, Dose 1 | 6
  Any Drowsiness, Dose 2: number analyzed (Participants) | 23
  Any Drowsiness, Dose 2 | 2
  Grade 3 Drowsiness, Dose 2: number analyzed (Participants) | 23
  Grade 3 Drowsiness, Dose 2 | 0
  Related Drowsiness, Dose 2: number analyzed (Participants) | 23
  Related Drowsiness, Dose 2 | 2
  Any Irritability, Dose 2: number analyzed (Participants) | 23
  Any Irritability, Dose 2 | 7
  Grade 3 Irritability, Dose 2: number analyzed (Participants) | 23
  Grade 3 Irritability, Dose 2 | 0
  Related Irritability, Dose 2: number analyzed (Participants) | 23
  Related Irritability, Dose 2 | 6
  Any Loss of appetite, Dose 2: number analyzed (Participants) | 23
  Any Loss of appetite, Dose 2 | 4
  Grade 3 Loss of appetite, Dose 2: number analyzed (Participants) | 23
  Grade 3 Loss of appetite, Dose 2 | 0
  Related Loss of appetite, Dose 2: number analyzed (Participants) | 23
  Related Loss of appetite, Dose 2 | 3
  Any Fever, Dose 2: number analyzed (Participants) | 23
  Any Fever, Dose 2 | 3
  Grade 3 Fever, Dose 2: number analyzed (Participants) | 23
  Grade 3 Fever, Dose 2 | 0
  Related Fever, Dose 2: number analyzed (Participants) | 23
  Related Fever, Dose 2 | 3
  Any Drowsiness, Dose 3: number analyzed (Participants) | 23
  Any Drowsiness, Dose 3 | 3
  Grade 3 Drowsiness, Dose 3: number analyzed (Participants) | 23
  Grade 3 Drowsiness, Dose 3 | 0
  Related Drowsiness, Dose 3: number analyzed (Participants) | 23
  Related Drowsiness, Dose 3 | 1
  Any Irritability, Dose 3: number analyzed (Participants) | 23
  Any Irritability, Dose 3 | 7
  Grade 3 Irritability, Dose 3: number analyzed (Participants) | 23
  Grade 3 Irritability, Dose 3 | 2
  Related Irritability, Dose 3: number analyzed (Participants) | 23
  Related Irritability, Dose 3 | 3
  Any Loss of appetite, Dose 3: number analyzed (Participants) | 23
  Any Loss of appetite, Dose 3 | 6
  Grade 3 Loss of appetite, Dose 3: number analyzed (Participants) | 23
  Grade 3 Loss of appetite, Dose 3 | 0
  Related Loss of appetite, Dose 3: number analyzed (Participants) | 23
  Related Loss of appetite, Dose 3 | 3
  Any Fever, Dose 3: number analyzed (Participants) | 23
  Any Fever, Dose 3 | 4
  Grade 3 Fever, Dose 3: number analyzed (Participants) | 23
  Grade 3 Fever, Dose 3 | 0
  Related Fever, Dose 3: number analyzed (Participants) | 23
  Related Fever, Dose 3 | 2
  Any Drowsiness, Across doses | 8
  Grade 3 Drowsiness, Across doses | 0
  Related Drowsiness, Across doses | 8
  Any Irritability, Across doses | 14
  Grade 3 Irritability, Across doses | 2
  Related Irritability, Across doses | 12
  Any Loss of appetite, Across doses | 9
  Grade 3 Loss of appetite, Across doses | 0
  Related Loss of appetite, Across doses | 8
  Any Fever, Across doses | 12
  Grade 3 Fever, Across doses | 0
  Related Fever, Across doses | 9

3. Primary Outcome: Number of Subjects Reporting Unsolicited Adverse Events (AEs)
Description: Unsolicited AE covers any AE reported in addition to those solicited during the clinical study and any solicited symptom with onset outside the specified period of follow-up for solicited symptoms. Any = occurrence of any unsolicited symptom regardless of intensity grade or relation to vaccination.
Time Frame: During the 31-days follow-up period after each dose of the study vaccine.
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | IPV Group
Number analyzed (Participants) | 25
Participants | 15

4. Primary Outcome: Number of Subjects Reporting Serious Adverse Events (SAEs)
Description: SAEs assessed included any untoward medical occurrence that resulted in death, was life-threatening, required hospitalization or prolongation of existing hospitalization, resulted in disability/incapacity or was a congenital anomaly/birth defect in the offspring of a study subject.
Time Frame: During the entire study period (from Dose 1 up to one month following last vaccine dose).
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | IPV Group
Number analyzed (Participants) | 25
Participants | 0

ADVERSE EVENTS:
Time Frame: Solicited symptoms: during the 4-day post-vaccination period after each vaccine dose. Unsolicited AEs: during the 31-day post-vaccination period after each vaccine dose. SAEs: during the entire study period (from Dose 1 up to one month following last vaccine dose).
Arm/Group | IPV Group
All-Cause Mortality (participants affected / at risk) | 0/25
Serious Adverse Events (participants affected / at risk) | 0/25
Other Adverse Events (participants affected / at risk) | 20/25
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | IPV Group (N=25)
Abdominal distension (Gastrointestinal disorders) | 1 (1)
Bronchitis (Infections and infestations) | 1 (1)
Conjunctivitis (Eye disorders) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 9 (17)
Diarrhoea (Gastrointestinal disorders) | 5 (7)
Dyspepsia (Gastrointestinal disorders) | 3 (4)
Erythema (Skin and subcutaneous tissue disorders) | 2 (3)
Irritability (Psychiatric disorders) | 14 (24)
Nasopharyngitis (Infections and infestations) | 4 (9)
Pain (General disorders) | 3 (4)
Pyrexia (General disorders) | 16 (21)
Skin infection (Infections and infestations) | 1 (1)
Somnolence (Nervous system disorders) | 8 (12)
Swelling (General disorders) | 2 (2)
Upper respiratory tract infection (Infections and infestations) | 7 (8)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.